CLINICAL TRIAL: NCT02949050
Title: Corn Based Occupational Rhinitis; SCIT Efficacy Study
Brief Title: Corn Occupational Rhinitis SCIT Efficacy Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: United Allergy Services (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Corn SCIT study-1
Record Dates: First submitted 2016-08-29; First posted 2016-10-31 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2017-10

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Experimental): the treatment -patients underwent SCIT and antihistamine/nasal steroid/use.
  Interventions: Biological: subcutaneous allergen immunotherapy (SCIT); Biological: SCIT
- Control Group (No Intervention): Control patient group only used antihistamines/nasal steroids but no SCIT

INTERVENTIONS:
Biological: subcutaneous allergen immunotherapy (SCIT) — 20 patients who (prior to study enrollment and initiation) completed more than 1 year of timothy grass SCIT vs. 20 control patients who underwent corn pollen exposure for for greater than one year during the same prestudy time interval. Efficacy will be assessed by analyses of symptom score surveys and quality of life surveys.
  Arms: Treatment Group
Biological: SCIT — Treatment group consists of patients who completed > 1 year of SCIT while control group patients did not undergo SCIT
  Arms: Treatment Group

SUMMARY:
Patients demonstrated allergic to corn pollen and timothy grass pollen (by allergy testing) who have undergone 1 to 2 years of subcutaneous allergen immunotherapy (SCIT) containing timothy grass extract with moderate symptomology (as documented via rhinitis symptom score surveys) will constitute the treatment group. Those who previously chose not to undergo SCIT who have documented symptomology and are skin test positive to corn pollen will constitute the control group. Prospective symptom score analyses and retrospective quality of life assessments (RQLQ) will be the primary and secondary efficacy outcome measures.

DETAILED DESCRIPTION:
Statistical assessment suggests enrollment of 20 patients into the treatment group (defined above) and an additional 20 into the control group. Patients will be matched for the level of symptomology (based on symptom score surveys) and residing/working on corn-crop farms. The premise for this study is the cross-reactivity of putative immunogenic sites between timothy grass pollen and corn pollen. based on consensus genetic sequences. Thus, the hypothesis is the use of Timothy grass extract containing immunotherapy would diminish symptomology to corn-based occupational rhinitis. Enrolled patients will have signed IRB approved consent forms and have undergone SCIT for 1 to 2 plus years (treatment group) or not undergone SCIT therapy for the same time period (control group). Potential contribution to symptom scores from other sources (e.g. Ragweed) will be analyzed by assessment of local pollen counts.Efficacy assessment will compare prospective symptom score results and retrospective quality of life survey scores between the treatment and control group responses.

ELIGIBILITY:
Inclusion Criteria for treatment group:

1. Completing more than 1 year of timothy grass SCIT
2. Residing/working on/near a corn farm
3. Having an initial symptom score value of > 8 (out of a possible 21).

Inclusion Criteria for control group:

1. Never treated with SCIT.
2. Residing/working on/near a corn farm
3. Having an initial symptom score value of > 8 (out of a possible 21).

All accepted enrolled patients are healthy volunteers.

Exclusion Criteria:

1. Negative allergy test to corn pollen,
2. Not residing on/near farm growing corn,
3. An initial symptom score of < 9.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Corn based Occupational Rhinitis symptom and medication score surveys | prior to study enrollment patients completed more than 1 year of SCIT. Actual study is 1 day to complete surveys.
  The completed symptom and medication score surveys will be contrasted from before to after therapy and between treatment and control groups.

SECONDARY OUTCOMES:
Corn based Occupational Rhinitis quality of life surveys | Actual survey completions take less than 1 day.
  secondary outcome measure-completed quality of life surveys will be assessed from before to after therapy and between the treatment and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: frederick m schaffer, md, Principal Investigator — United Allergy Services

IPD SHARING:
Plan to Share IPD: No